CLINICAL TRIAL: NCT01721694
Title: Association of Azithromycin 1,5%/Loteprednol 0,5% Eye Drops Versus Individual Administration of Azithromycin 1,5% and Loteprednol 0,5% in the Treatment of Ocular Inflammation and Infection
Brief Title: Antibiotic Steroid Combination Compared With Individual Administration in the in the Treatment of Ocular Inflammation and Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn by industry
Sponsor: Adapt Produtos Oftalmológicos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZILOT-12; 131.835 (Other: CEP-UNIFESP-Plataforma Brasil)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Ocular Inflammation; Infection Associated Blepharitis; Keratitis; Conjunctivitis, Bacterial
Keywords: bacterial ocular inflammation; blepharitis; keratitis; conjunctivitis
MeSH Terms: conditions — Keratitis; Conjunctivitis, Bacterial; Blepharitis; Conjunctivitis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- azithromycin 1.5%/Loteprednol 0,5% + placebo (Experimental): fixed combination of azithromycin 1.5% / Loteprednol 0,5% eye drops + placebo eye drops
  Interventions: Drug: azithromycin 1.5%/Loteprednol 0,5% + placebo
- azithromycin 1.5% + Loteprednol 0,5% (separately) (Active Comparator): azithromycin 1.5% + Loteprednol 0,5% eye drops (separately)
  Interventions: Drug: azithromycin 1.5% + Loteprednol 0,5% (separately)

INTERVENTIONS:
Drug: azithromycin 1.5%/Loteprednol 0,5% + placebo — 1 drop, AO, QID
  Arms: azithromycin 1.5%/Loteprednol 0,5% + placebo
Drug: azithromycin 1.5% + Loteprednol 0,5% (separately) — 1 drop, QID, AO
  Other Names: azithromycin 1.5% + Loteprednol 0,5% eye drops (separately)
  Arms: azithromycin 1.5% + Loteprednol 0,5% (separately)

SUMMARY:
To evaluate the efficacy and safety of fixed combination of azithromycin 1.5% + 0.5% Loteprednol eye drops for the treatment of ocular inflammation and infection associated bacterial blepharitis and / or keratitis and / or conjunctivitis compared with the individual administration of azithromycin 1.5% and 0.5% Loteprednol (separately).

DETAILED DESCRIPTION:
Estimated to be admitted a total of approximately 60 patients showing blepharitis and / or keratitis and / or conjunctivitis: 30 patients will be assigned to the group of Azithromycin 1.5%/Loteprednol 0.5% Eye Drops (fixed combination) + placebo and 30 patients will be assigned to the group of Azithromycin 1.5% + 0.5% Loteprednol (separately)

ELIGIBILITY:
Inclusion Criteria:

* Patients were male or female, of any race and age minimum of 18 years.
* Blepharitis should provide diagnostic and / or keratitis and / or conjunctivitis with or without bacterial involvement corneal by biomicroscopy, with positive staining corneal fluorescein and also provide a composite score ≥ 2 on: bulbar conjunctival hyperemia, eyelid conjunctiva, secretion / exudate conjunctival erythema and flaking eyelids / eyelid crust on at least one eye (the same eye) on Day 1 visit

Exclusion Criteria:

* Intraocular hypertension or uncontrolled glaucoma.
* Use of contact lenses during the study.
* Capacity unilateral visual only.
* Suspected fungal infection, viral (eg, herpes simplex epithelial, dendritic keratitis) or Acanthamoeba, or any other disease where the use of corticosteroids is contraindicated.
* Use of any topical ophthalmic medications preserved during study participation. Not be allowed eyedrops preserved (eg artificial tears).
* Use of any antibacterial agent oral or topical ophthalmic until 72 hours prior to study entry.
* Use of systemic steroids within 14 days prior to study entry. Ophthalmic topical steroids or nonsteroidal anti-inflammatory drugs (NSAIDs), until one week before admission to the study. Will not be allowed to use these medications during study participation. Will not be allowed to use nasal steroids during the study. Will be allowed to use inhaled steroids to aid inhaler. Will be allowed steroids dermal topics.
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) systemic up to 24 hours prior to study entry or at any time during the study, unless the patient is under treatment regimen with stable (not necessary) for at least 2 months before Admission and therapy continues throughout the study.
* Any disturbance or ocular or systemic disease, complicating factors or structural abnormality that affects the conduct or outcome of the study in a negative way or represents an undue risk to patient safety, according to the opinion of the investigator.
* Any current immunosuppressive disorder (eg, HIV-positive), or immunosuppressive therapy (including chemotherapy).
* Known allergy or suspected allergy or hypersensitivity to fluoroquinolones, to steroids or any other component of the study drug;
* Pregnant or lactating. (Women of childbearing age may be admitted if they use contraception and submit urine pregnancy test negative);
* Any patient who has a family member who participates in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | Day 8
  Clinical cure achieved when the score of the cardinal ocular signs (hyperemia in the bulbar conjunctiva, palpebral, exudate / conjunctival discharge, eyelid erythema and flaking / crust eyelid) is zero at the time of conclusion of the study (D8)

SECONDARY OUTCOMES:
irradication of pathogens | Day 8
  Success obtained with microbiological irradication of pathogens present at baseline

OTHER OUTCOMES:
ophthalmic evaluation | Day 4 and Day 8
  decrease of visual acuity, corneal/anterior chamber changes, IOP increase and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr., MD, Principal Investigator — Federal University of São Paulo / Hospital São Paulo
Locations (1):
- Department of Ophthalmology of Hospital São Paulo, São Paulo, São Paulo, Brazil